CLINICAL TRIAL: NCT00132899
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Multi-Centre Study to Evaluate the Safety and Efficacy of Infliximab in Combination With Methotrexate for the Long-term Treatment of Crohn's Disease (CD)
Brief Title: COMMIT (Combination Of Maintenance Methotrexate-Infliximab Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP0401
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2005-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; multi-centre randomized placebo-controlled; infliximab; methotrexate; inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Active Comparator): Methotrexate and infliximab combination
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo plus infliximab combination
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate and infliximab combination
  Arms: Methotrexate
Drug: Placebo — Placebo and infliximab combination therapy.
  Arms: Placebo

SUMMARY:
The primary objective is to compare the efficacy and safety of infliximab plus methotrexate to infliximab alone for the long-term control of signs and symptoms of Crohn's disease (CD) in patients with symptoms that are persistent enough to require corticosteroid therapy.

DETAILED DESCRIPTION:
The current approach to the treatment of Crohn's Disease is based on "step care". This strategy is relatively ineffective for the long-term management of patients who require treatment with corticosteroids. Although azathioprine, methotrexate and infliximab are modestly effective in this high-risk population, long-term corticosteroid-free response rates are low. Thus combination therapy is an attractive option to explore. Based on a favourable experience with dual therapy in the treatment of rheumatoid arthritis and the demonstrated efficacy of methotrexate in corticosteroid-dependent CD, we expect that combination therapy with methotrexate and infliximab will be significantly more effective than infliximab monotherapy. Furthermore combined therapy is likely to be highly effective in preventing formation of the antibodies to infliximab that are an important limitation to the continued successful use of this drug.

This is a randomized, placebo-controlled, double-blind, parallel group, multi-centre study. Subjects who have initiated corticosteroid induction therapy within the preceding 6 weeks will be randomized (irrespective of CDAI defined disease activity) in a 1:1 ratio to either methotrexate or placebo for a period of 50 weeks in combination with infliximab administered for 8 infusions. Randomization will be stratified by:

* Treatment with or without Imuran/6-mercaptopurine in the 2-12 months prior to randomization;
* Prednisone dose <20 mg or ≥20 mg daily at randomization;
* CDAI <150 or ≥150 at randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male, or non-pregnant/non-lactating females, 18 or older
* Established Crohn's disease with active symptoms requiring prednisone therapy.
* Females of child-bearing potential must have a negative pregnancy test and must agree to use adequate contraception

Exclusion Criteria:

* Intolerance or hypersensitivity to infliximab, methotrexate, prednisone and or known allergy to murine proteins or other chimeric proteins
* Are pregnant, nursing, or planning pregnancy (both men and women) during or in the 6 months after the study
* In the 2 months prior to screening, have had a serious infection, or have been hospitalized for and/or treated with intravenous (IV) antibiotics for infection. In the 6 months prior to screening, have had an opportunistic infection.
* After screening, need to continue non-study medical therapy for CD
* In the 8 weeks prior to screening, have received any of the following: systemic steroid therapy, azathioprine, 6-mercaptopurine, cyclosporine, probiotic products, or omega-3 fatty acids
* Have received any of the following: biologics in the last 6 months; methotrexate in the last year; and/or ever received infliximab.
* Have any of the following: biopsy-proven cirrhosis, clinically important lung disease, pre-existing demyelinating disorder, systemic lupus erythematosus, congestive heart failure, diabetes mellitus (insulin dependent), increased risk for steroid-related side effects, body weight 40% higher than standard, human immunodeficiency virus and/or hepatitis B or hepatitis C
* Have any of the following: an active draining fistula as the primary manifestation of CD; documented short bowel syndrome; a stoma; or severe, and/or fixed symptomatic stenosis of the intestine.
* Have had any of the following: clinically important bowel obstruction in the last 3 months; a bowel resection in the last 3 months; and/or other intra-abdominal surgery within 6 months.
* Clinically significant impairment in cardiac, liver or renal function; central nervous system (CNS), pulmonary, hematological, immunological, vascular and gastrointestinal disease in addition to CD; current malignancy or malignancy within 5 years prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Treatment success as defined by the proportion of subjects in clinical remission (i.e. complete discontinuation of prednisone therapy and a CDAI score of <150) at week 14, and maintenance of clinical remission between study weeks 14 and 50 | one year

SECONDARY OUTCOMES:
Efficacy of infliximab therapy in combination with methotrexate on disease activity using the Crohn's Disease Activity Index (CDAI) and Investigator and Subject Global Ratings | one year
Effects of infliximab therapy in combination with methotrexate on health-related quality of life | one year
Proportion of subjects who develop antibodies to infliximab | one year

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Feagan, MD, M.Sc, Study Director — Robarts Clinical Trials, Robarts Research Institute
Locations (1):
- Robarts Clinical Trials, Robarts Research Institute, London, Ontario, Canada

REFERENCES:
- [Background] Bernstein CN, Blanchard JF, Rawsthorne P, Wajda A. Epidemiology of Crohn's disease and ulcerative colitis in a central Canadian province: a population-based study. Am J Epidemiol. 1999 May 15;149(10):916-24. doi: 10.1093/oxfordjournals.aje.a009735. PMID 10342800
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078
- [Background] Munkholm P, Langholz E, Davidsen M, Binder V. Disease activity courses in a regional cohort of Crohn's disease patients. Scand J Gastroenterol. 1995 Jul;30(7):699-706. doi: 10.3109/00365529509096316. PMID 7481535
- [Derived] Feagan BG, McDonald JW, Panaccione R, Enns RA, Bernstein CN, Ponich TP, Bourdages R, Macintosh DG, Dallaire C, Cohen A, Fedorak RN, Pare P, Bitton A, Saibil F, Anderson F, Donner A, Wong CJ, Zou G, Vandervoort MK, Hopkins M, Greenberg GR. Methotrexate in combination with infliximab is no more effective than infliximab alone in patients with Crohn's disease. Gastroenterology. 2014 Mar;146(3):681-688.e1. doi: 10.1053/j.gastro.2013.11.024. Epub 2013 Nov 21. PMID 24269926